

### - Sistema Socio Sanitario



Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

#### STUDY PROTOCOL

The Italian REgistry of pulmonary Non-tuberculous mycobactEria – IRENE

Version #: 2.0

Date: June 21st, 2017

Sistema Socio Sanitario





Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

U.O.S Fibrosi Cistica Sez. Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

**Study Sponsor:** 

UO di Broncopneumologia, Dipartimento delle Units multispecialistiche e dei trapianti / Area

Cardio-Polmonare, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milano

**Principal Investigator:** 

Prof. Stefano Aliberti, Dipartimento di Fisiopatologia Medico-Chirurgica e dei Trapianti,

Università degli Studi di Milano, UO di Broncopneumologia, Dipartimento delle Units

multispecialistiche e dei trapianti / Area Cardio-Polmonare, Fondazione IRCCS Ca' Granda

Ospedale Maggiore Policlinico, Milano; E-mail: stefano.aliberti@unimi.it.

**Executive committee:** 

Prof. Stefano Aliberti, Dipartimento di Fisiopatologia Medico-Chirurgica e dei Trapianti,

Università degli Studi di Milano, UO di Broncopneumologia, Dipartimento delle Units

multispecialistiche e dei trapianti / Area Cardio-Polmonare, Fondazione IRCCS Ca' Granda

Ospedale Maggiore Policlinico, Milano; E-mail: stefano.aliberti@unimi.it.

Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico

Sistema Socio Sanitario



Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: <u>broncopneumologia@policlinico.mi.it</u>

U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

Prof. Francesco Blasi, Dipartimento di Fisiopatologia Medico-Chirurgica e dei Trapianti,
 Università degli Studi di Milano, UO di Broncopneumologia, Dipartimento delle Units
 multispecialistiche e dei trapianti / Area Cardio-Polmonare, Fondazione IRCCS Ca' Granda

Ospedale Maggiore Policlinico, Milano; E-mail: francesco.blasi@unimi.it.

• Dr. Luigi Ruffo Codecasa, Centro regionale di riferimento per TB, Istituto Villa Marelli, ASST

Grande Ospedale Metropolitano Niguarda, Milano; E-mail:

luigiruffo.codecasa@ospedaleniguarda.it

Prof. Andrea Gori, Scuola di Medicina e Chirurgia, Università degli Studi di Milano Bicocca,

UO Malattie Infettive, ASST di Monza, Ospedale San Gerardo, Monza; E-Mail:

andrea.gori@unimib.it

**Scientific Committee** 

1. Prof. Stefano Aliberti, Dipartimento di Fisiopatologia Medico-Chirurgica e dei Trapianti,

Università degli Studi di Milano, UO di Broncopneumologia, Dipartimento delle Units

multispecialistiche e dei trapianti / Area Cardio-Polmonare, Fondazione IRCCS Ca' Granda

Ospedale Maggiore Policlinico, Milano





Sistema Socio Sanitario



Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

U.O.S Fibrosi Cistica Sez. Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

2. Prof. Francesco Blasi, Dipartimento di Fisiopatologia Medico-Chirurgica e dei Trapianti, Università degli Studi di Milano, UO di Broncopneumologia, Dipartimento delle Units multispecialistiche e dei trapianti / Area Cardio-Polmonare, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milano

3. Dr. Luigi Ruffo Codecasa, Centro regionale di riferimento per TB, Istituto Villa Marelli, ASST Grande Ospedale Metropolitano Niguarda, Milano

4. Prof. Andrea Gori, Scuola di Medicina e Chirurgia, Università degli Studi di Milano Bicocca, UO Malattie Infettive, ASST di Monza, Ospedale San Gerardo, Monza

5. Prof. Giovanni Sotgiu, Clinical Epidemiology and Medical Statistics Unit, Department of Biomedical Sciences, Università degli Studi di Sassari, Sassari, Italia

6. Dr Stefano Nardini, UO di Pneumotisiologia, Ospedale di Vittorio Veneto, Treviso, Italia

Dr Mehdi Mirsaeidi, Division of Pulmonary and Critical Care, University of Miami, 1600 NW,
 Miami, FL 33136, USA; Miami VA Medical Center, 1201 N.W. 16th St., Miami, FL 33125,
 USA.

8. Dr Enrico Tortoli, Emerging Bacterial Pathogens Unit, IRCCS Ospedale San Raffaele, Milano, Italia

9. Dr Giorgio Besozzi, Stop TB Italia, Milano, Italia











Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: <u>broncopneumologia@policlinico.mi.it</u>

U.O.S Fibrosi Cistica Sez. Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

10. Dr Alberto Matteelli, Clinic of Infectious and Tropical Diseases, University of Brescia and Brescia Spedali Civili General Hospital, WHO Collaborating Centre for TB/HIV and TB Elimination, Brescia, Italia

- 11. Dr Antonio Di Biagio, IRCCS-AOU-San Martino-IST, Infectious Disease Clinic, Genova, Italia
- 12. Dr Andrea Calcagno, Università degli Studi di Torino
- 13. Dr Girardi Spallanzani, UOC Epidemiologia Clinica Dipartimento di Epidemiologia e Ricerca Preclinica, Clinical Epidemiology Unit Department of Epidemiology and Preclinical Research Istituto Nazionale Malattie Infettive "L. Spallanzani" IRCCS Via Portuense 292, 00149 Roma
- 14. Dr Giuliana Previdi, rappresentate pazienti
- 15. Dr Baroukh Maurice Assael, Università degli Studi di Milano, UO di Broncopneumologia, Dipartimento delle Units multispecialistiche e dei trapianti / Area Cardio-Polmonare, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milano





### - Sistema Socio Sanitario



Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: <u>broncopneumologia@policlinico.mi.it</u>

U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>



Sistema Socio Sanitario



Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

**BACKGROUND** 

Pulmonary disease due to non-tuberculous mycobacteria (NTM) has always been a tangible clinical entity [1]. An increase in NTM pulmonary and extra-pulmonary morbidity and mortality has been documented in Italy and worldwide, especially among patients suffering from chronic respiratory diseases, including bronchiectasis, chronic obstructive pulmonary disease (COPD), or cystic fibrosis (CF), as well as among HIV-positive and other immunocompromised patients [2-11]. Several determinants of the increasing epidemiological trend have been identified: the aging of the population with high prevalence of chronic and debilitating diseases; an intensified use of immunosuppressive therapies; a broader use of chest CT; a high diagnostic yield of microbiological conventional and molecular techniques; an increasing environmental exposure to NTM; an increase use of antibiotics which can favor the occurrence of niches for NTM; declining rates of *M. tuberculosis* infection; and a potential impact of person-to-person transmission as recently suggested among CF patients [12,13].

The epidemiology of patients suffering from a pulmonary disease due to NTM (NTM-PD), which is characterized by symptomatic, progressive inflammatory lung damage and defined in 2007 in the ATS/IDSA guidelines, still remains unclear [14,15]. Epidemiological and clinical uncertainties on NTM-PD cause significant confusion for clinicians in daily clinical practice when asked to diagnose







Dipartimento delle Units multispecialistiche e dei Trapianti - Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: <u>broncopneumologia@policlinico.mi.it</u>

U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

NTM-PD. The clinical relevance of NTM respiratory infections significantly varies from patient to patient, and the interplay between exposure- and host-related factors is poorly understood [15]. NTM-PD shows a wide spectrum of clinical manifestations and frequently is diagnosed in the context of concomitant respiratory diseases (e.g., bronchiectasis or CF) [3]. Geographical diversity is another important factor in the epidemiology of NTM. A large inter- and intra-country heterogeneity in distribution of NTM species has been recently shown [16,17]. Finally, an Italian experience described NTM-PD risk factors whose qualitative and quantitative ascertainment could help clinicians to discriminate between colonization and disease [18].

Reporting of NTM-PD to health authorities is often not mandated in several countries and the current estimates have been obtained from sentinel surveillance or laboratory-based studies, retrospective cohort studies, or audits of administrative databases. Only a few European countries (*i.e.*, UK, Greece, Germany, and the Netherlands) have provided epidemiological data, showing an incidence rate of NTM isolation ranging from 2.9 to 7.0 per 100,000 population and a NTM-PD prevalence of 0.7-1.7 per 100,000 population [19-21]. Until now no data have been published on the epidemiology of respiratory NTM infections in Italy.

On this basis, robust national longitudinal data are needed. This manuscript describes the protocol of the first Italian registry of adult patients with respiratory infections caused by NTM.







Sistema Socio Sanitario



Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

METHODOLOGY OF THE IRENE REGISTRY

Study design

The Italian registry of pulmonary NTM (IRENE) is an observational, multicenter, prospective, cohort study enrolling consecutive adult patients with either a NTM respiratory infection or NTM-PD. The coordinating center is located at the Pulmonary Department of the Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (hereby referred to as Policlinico Hospital), Milan, Italy, where the central approval from the Ethical Committee (EC) for this study was obtained on March 6<sup>th</sup>, 2017, and the first patient was enrolled on April 21<sup>st</sup>, 2017. A total of 35 centers, including mainly pulmonary and infectious disease (ID) departments, requested to join the registry, see Figure 1. All the centers are required to obtain local EC approval before entering the registry. Additionally, other EC approvals will be required by IRENE centers prior to commencement of the study at each site. All patients must provide written informed consent to participate in the registry. The study is sponsored by the Policlinico Hospital in Milan.

– Sistema Socio Sanitario





Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

Study subjects

Adult (≥18 years) patients with all of the following will be included in the registry: 1) at least one positive culture for any NTM species from any respiratory sample; 2) at least one positive culture for NTM isolated in the year prior the enrolment and/or prescribed NTM treatment in the year prior the enrolment; 3) Given consent to inclusion in the study. No exclusion criteria are applied to the study in order to increase the generalizability of the results. The inclusion criteria of the registry clearly identify a population of patients characterized by a recent/ongoing history of either a NTM infection or NTM-PD. The IRENE Steering Committee decided not to limit the enrolment to patients with NTM-PD, but to follow up also patients with a recent NTM infection not fulfilling the 2007 ATS/IDSA criteria for NTM-PD [15].

Patients included in the registry are mainly recruited among pulmonary and ID out- and in-patient services. Adult CF, lung transplant, and tuberculosis clinics represent other recruitment centers. A heterogeneous population of patients with NTM infection/NTM-PD sharing different clinical



Sistema Socio Sanitario



Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

phenotypes is expected to be enrolled in the registry. IRENE has a special focus on four patients' categories: 1) immunocompetent/bronchiectatic, 2) HIV-positive, 3) CF and 4) lung transplanted patients. 500 patients are expected to be enrolled in the registry by the end of 2020. The registry has been developed to accept an unlimited number of patients and no deadlines have been decided.

Data Collection, definitions and quality control

Patients are managed according to standard operating procedures (SOPs) implemented in each IRENE clinical center without any interference from the study team. A baseline case report form (CRF) is collected at patient's enrolment including demographics, comorbidities, microbiological, laboratory, functional, radiological, clinical, and treatment data. Then, study investigators will enter follow-up data on an annual basis, see online supplement. Furthermore, a "start treatment" and a "stop treatment" CRF will also be collected. The database incorporates automated logic checks put in place to avoid the collection of out-of-range values. Once the case is entered into the registry, two members of the study team (SA and MS) manually verified its consistency and data queries will be solved with the local study investigator. In case of unresolved queries or incomplete cases, they will be rejected to have high quality data. To assure the high quality of the data, random audit will also be conducted at study sites.

Sistema Socio Sanitario

Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico



Dipartimento delle Units multispecialistiche e dei Trapianti - Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

U.O.S Fibrosi Cistica Sez. Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

**IRENE Biobank** 

An IRENE biobank has also been developed within the network and linked to the clinical data of the registry. IRENE sites can collect samples, including blood, serum, plasma, respiratory specimens (e.g., sputum, induced sputum, tracheal aspirate, or bronchoalveolar lavage), urine, and NTM isolates at the first visit and during follow up on a voluntary basis. The same SOPs for biological collection, processing, and storage (first locally and then centralized at the Policlinico Hospital in Milan for analysis) will be adopted by all IRENE sites.

The registry governance and the IRENE network

The registry is held securely at the Health Informatics Centre (HIC) of the Policlinico Hospital in Milan, Italy, and de-identified data will be accessible to the study investigators; however, they can have unrestricted access to their own data. Analysis of the entire IRENE database will be allowed after the submission of a specific research question, along with a complete study protocol, to the IRENE Executive Committee. The database will be run in accordance with the principles of Good Clinical Practice. Study results will be disseminated in the form of annual reports, conference

Sistema Socio Sanitario





Dipartimento delle Units multispecialistiche e dei Trapianti - Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

abstracts, and peer reviewed publications. The IRENE network will follow the International Committee of Medical Journal Editors recommendations regarding authorship.

IRENE is the official Italian network within the EMBARC European NTM registry [22]. All Italian patients included in the European NTM registry will be enrolled through IRENE and IRENE data will be incorporated into the European NTM registry.

IRENE also promotes multi-disciplinary education and patient-professional collaboration in the field of NTM through its relationship with national scientific societies. So far, IRENE received the endorsement by the Italian Respiratory Society (IRS/SIP), the Italian Society of Cystic fibrosis and STOP TB Italia, with pending endorsement from other national scientific societies. There is a lack of a platform for communication between patients with NTM infection/NTM-PD and physicians in Italy and some patients within the IRENE network already expressed their will to develop a patient advisory group.







Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

#### **REFERENCES**

- 1. Piersimoni C, Scarparo C. Pulmonary infections associated with non-tuberculous mycobacteria in immunocompetent patients. Lancet Infect Dis. 2008 May;8(5):323-34
- 2. Rindi L, Garzelli C. Increase in non-tuberculous mycobacteria isolated from humans in Tuscany, Italy, from 2004 to 2014. BMC Infect Dis. 2016 Feb 1;16:44
- 3. Bonaiti G, Pesci A, Marruchella A, Lapadula G, Gori A, Aliberti S. <u>Nontuberculous</u>

  Mycobacteria in Noncystic Fibrosis Bronchiectasis. Biomed Res Int. 2015;2015:197950.
- 4. Faverio P, Stainer A, Bonaiti G, Zucchetti SC, Simonetta E, Lapadula G, Marruchella A, Gori A, Blasi F, Codecasa L, Pesci A, Chalmers JD, Loebinger MR, Aliberti S. Characterizing Non-Tuberculous Mycobacteria Infection in Bronchiectasis. Int J Mol Sci. 2016 Nov 16;17
- 5. Kendall BA, Winthrop KL. Update on the epidemiology of pulmonary nontuberculous mycobacterial infections. Semin Respir Crit Care Med 2013;34:87–94
- 6. Prevots DR, Marras TK. Epidemiology of human pulmonary infection with nontuberculous mycobacteria: a review. Clinics in Chest medicine 2015; 36 (1): 13-34





Sistema Socio Sanitario





Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

- 7. van der Werf MJ, Ködmön C, Katalinić-Janković V, Kummik T, Soini H, Richter E, et al. Inventory study of non-tuberculous mycobacteria in the European Union. BMC Infect Dis. 2014;14:62.
- 8. Ringshausen FC, Apel RM, Bange FC, de Roux A, Pletz MW, Rademacher J, et al. Burden and trends of hospitalisations associated with pulmonary non- tuberculous mycobacterial infections in Germany, 2005–2011. BMC Infect Dis. 2013;13:231.
- 9. Moore JE, Kruijshaar ME, Ormerod LP, Drobniewski F, Abubakar I. Increasing reports of non-tuberculous mycobacteria in England, Wales and Northern Ireland, 1995–2006. BMC Public Health. 2010;10:612.
- 10. Biondi G, Sotgiu G, Dore S, Molicotti P, Ruggeri M, Aliberti S, Satta R. <u>Beyond pulmonary</u> nontuberculous mycobacteria disease: do extra-pulmonary forms represent an emerging <u>clinical and public health threat?</u> ERJ Open Res. 2017 Sep 19;3(3). pii: 00091-2017
- 11. Mirsaeidi M, Machado RF, Garcia JG, Schraufnagel DE. Nontuberculous mycobacterial disease mortality in the united states, 1999-2010: A population-based comparative study. PLoS One 2014;9(3):e91879
- 12. Brode SK, Daley CL, Marras TK. The epidemiologic relationship between tuberculosis and non-tuberculous mycobactyerial disease: a systematic review. IJTLD 2014; 18 (11): 1370-7



Sistema Socio Sanitario



Dipartimento delle Units multispecialistiche e dei Trapianti - Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

13. Bryant CE; Grogono DM, Rodriguez-rincon D. Population-level genomics identifies the emergence and global spread of a human transmissible multidrug-resistant nontuberculuous mycobacterium. Science 2016

14. Diel R, Jacob J, Lampenius N, Loebinger M, Nienhaus A, Rabe KF, Ringshausen FC. <u>Burden of non-tuberculous mycobacterial pulmonary disease in Germany.</u> Eur Respir J. 2017 Apr 26;49(4)

15. Griffith DE, Aksamit T, Brown-Elliott BA, Catanzaro A, Daley C, Gordin F, Holland SM, Horsburgh R, Huitt G, Iademarco MF, Iseman M, Olivier K, Ruoss S, von Reyn CF, Wallace RJ Jr, Winthrop K; ATS Mycobacterial Diseases Subcommittee; American Thoracic Society; Infectious Disease Society of America. An official ATS/IDSA statement: diagnosis, treatment, and prevention of nontuberculous mycobacterial diseases. Am J Respir Crit Care Med. 2007 Feb 15;175(4):367-416. Review. No abstract available. Erratum in: Am J Respir Crit Care Med. 2007 Apr 1;175(7):744-5.

16. Hoefsloot W, van Ingen J, Andrejak C, Angeby K, Bauriaud R, Bemer P, et al. The geographic diversity of nontuberculous mycobacteria isolated from pulmonary samples: an NTM-NET collaborative study. Eur Respir J 2013;42:1604–13







Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: <u>broncopneumologia@policlinico.mi.it</u>

U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

17. Mirsaeidi M, Vu A, Leitman P, Sharifi A, Wisliceny S, Leitman A, Schmid A, Campos M, Falkinham J, Salathe M. A patient-based analysis of the geographic distribution of mycobacterium avium complex, mycobacterium abscessus, and mycobacterium kansasii infections in the united states. Chest 2017;151(4):947-950

18. Mencarini J, Cresci C, Simonetti MT, Truppa C, Camiciottoli G, Frilli ML, Rogasi PG, Veloci S, Pistolesi M, Rossolini GM, Bartoloni A, Bartalesi F. Non-tuberculous mycobacteria: epidemiological pattern in a reference laboratory and risk factors associated with pulmonary disease. Epidemiol Infect. 2017 Feb;145(3):515-522

19. Henry MT, Inamdar L, O'Riordain D, Schweiger M, Watson JP. Nontuberculous mycobacteria in non-HIV patients: epidemiology, treatment and response. Eur Respir J 2004;23:741–6

- 20. Gerogianni I, Papala M, Kostikas K, Petinaki E, Gourgoulianis KI. Epidemiology and clinical significance of mycobacterial respiratory infections in Central Greece. Int J Tuberc Lung Dis 2008;12:807–12
- 21. van Ingen J, Bendien SA, de Lange WC, Hoefsloot W, Dekhuijzen PN, Boeree MJ, et al.

  Clinical relevance of non-tuberculous mycobacteria isolated in the Nijmegen-Arnhem region, the Netherlands. Thorax 2009;64:502–6







Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: <u>broncopneumologia@policlinico.mi.it</u>

22. Chalmers JD, Aliberti S, Polverino E, Vendrell M, Crichton M, Loebinger M, Dimakou K, Clifton I, van der Eerden M, Rohde G, Murris-Espin M, Masefield S, Gerada E, Shteinberg M, Ringshausen F, Haworth C, Boersma W, Rademacher J, Hill AT, Aksamit T, O'Donnell A, Morgan L, Milenkovic B, Tramma L, Neves J, Menendez R, Paggiaro P, Botnaru V, Skrgat S, Wilson R, Goeminne P, De Soyza A, Welte T, Torres A, Elborn JS, Blasi F. The EMBARC European Bronchiectasis Registry: protocol for an international observational study. ERJ Open Res. 2016 Jan 20;2(1).

Figure 1. IRENE centers



# Sistema Socio Sanitario



Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

U.O.S Fibrosi Cistica Sez. Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

